CLINICAL TRIAL: NCT06696274
Title: Investigation of the Relationship Between Kinesiophobia and Pain, Balance, Quality of Life and Mental Status in Hemodialysis Patients
Brief Title: Kinesiophobia, Pain, Balance, Quality of Life and Mental Status in Hemodialysis Patients
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-12/101
Record Dates: First submitted 2024-11-06; First posted 2024-11-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hemodialysis; End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hemodialysis patients

SUMMARY:
The aim of our study was to investigate the relationship between kinesiophobia and pain, balance, physical performance, quality of life and mental status in patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease receiving hemodialysis
* Receiving hemodialysis for more than 3 months
* Being clinically stable
* Volunteering to participate in this stud

Exclusion Criteria:

-Having musculoskeletal disorders that may affect physical performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal disease receiving hemodialysis will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | Day 1
  It will be evaluated with the Tampa Kinesiophobia scale.The total score ranges from 17-68, with a score above 37 indicating a high degree of kinesiophobia.
Pain | Day 1
  Will be evaluated with a numeric rating scale. Higher scores indicate worse outcomes.
Balance | Day 1
  It will be assessed with a timed up and go test
Physical performance | Day 1
  It will be evaluated with five-repetition sit-to-stand test

SECONDARY OUTCOMES:
Quality of life | Day 1
  It will be evaluated with the Short Form-36 Quality of Life scale.The subscales rate health from 0 to 100, with 0 indicating poor health and 100 indicating good health.
Mental health | Day 1
  It will be assessed using the Hospital Anxiety and Depression scale. The lowest score they can get from both subscales is 0 and the highest score is 21.High scores indicate high levels of anxiety and depression
Comorbidity level | Day 1
  It will be evaluated with the Charlson Comorbidity Index. Total score is between 0-37. Higher scores indicate worse outcomes and higher risk of death.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Topal, Study Chair — Kirsehir Ahi Evran University; Aydin Guclu, Study Chair — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)